CLINICAL TRIAL: NCT07352059
Title: Safety and Efficacy of Midazolam Alone Versus Midazolam With Ketorolac in Patients Undergoing Flexible Bronchoscopy.
Brief Title: Midazolam Alone Versus Midazolam With Ketorolac for Sedation During Flexible Bronchoscopy.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SYED HAIDER ALI (Other Government)
Responsible Party: Sponsor-Investigator, SYED HAIDER ALI, Registrar, Services Institute of Medical Sciences, Pakistan
Organization: Services Institute of Medical Sciences, Pakistan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB/2025/1732/SIMS
Record Dates: First submitted 2026-01-05; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Sedation and Analgesia Management in Patients Undergoing Flexible Bronchoscopy
Keywords: Flexible bronchoscopy, midazolam, ketorolac, sedation, analgesia, patient comfort, safety, procedural tolerance
MeSH Terms: conditions — Agnosia | interventions — Midazolam; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Intervention Model Description: Randomized, controlled study comparing midazolam alone versus midazolam with ketorolac for sedation during flexible bronchoscopy. Adult patients will be assigned to one of the two groups. Primary outcomes: sedation quality, patient comfort, and procedure-related adverse events. Secondary outcomes: hemodynamic stability and recovery time. All drugs are approved and used in standard clinical practice. No investigational drugs are involved.
Masking Description: Not applicable. No parties are masked in this open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Midazolam Sedation Alone for Flexible Bronchoscopy (Active Comparator): Participants receive intravenous midazolam alone for procedural sedation during flexible bronchoscopy. Safety and efficacy outcomes will be measured.
  Interventions: Drug: Midazolam Alone
- Midazolam with Ketorolac Sedation for Flexible Bronchoscopy (Active Comparator): Participants receive intravenous midazolam combined with ketorolac for procedural sedation during flexible bronchoscopy. Safety and efficacy outcomes will be measured.
  Interventions: Drug: Midazolam + ketorolac

INTERVENTIONS:
Drug: Midazolam Alone — Intravenous midazolam 0.05 mg/kg (maximum 5 mg), administered in divided doses 2.5mg bolus followed by 1.5mg and 1mg bolus if required. Each midazolam dose will be followed by saline bolus of 10 ml to facilitate rapid drug delivery.
  Arms: Midazolam Sedation Alone for Flexible Bronchoscopy
Drug: Midazolam + ketorolac — Intravenous ketorolac 30 mg, will be administered 10-15 minutes before bronchoscopy. Intravenous midazolam 0.05 mg/kg (maximum 5 mg) administered in divided doses 2.5mg bolus followed by 1.5mg and 1mg bolus if required.
  Other Names: Dormicum; Toradol
  Arms: Midazolam with Ketorolac Sedation for Flexible Bronchoscopy

SUMMARY:
Flexible bronchoscopy has evolved into a vital diagnostic and therapeutic intervention in respiratory medicine due to its frequent and diverse applications. It enables direct visualization of the tracheobronchial tree and facilitates procedures such as bronchoalveolar lavage, tissue sampling, and foreign body extraction. However, despite its clinical importance, the procedure is associated with patient discomfort due to airway manipulation, hypoxia, coughing and procedural pain. These discomforts can lead to poor patient cooperation, excessive movement, procedure related anxiety and even premature termination of the procedure, consequently affecting diagnostic accuracy and patient safety.

Multiple technique has been used should be improved procedural tolerance and adequate sedation is of the prime importance. Sedation during bronchoscopy helps in reducing anxiety, suppressing the cough reflex, minimizing procedural duration and reduce overall complications. An ideal sedative agent should allow quick procedural recovery, ensuring patient comfort, procedural safety and overall diagnostic yield.

Sedative agents have dose dependent side effects including bradycardia, hypotension, respiratory depression, hypoxia which may lead to termination of procedure. Higher doses of topical analgesia with lignocaine can lead to seizures and bradycardia.

Multiple studies elaborate that addition of analgesia with some dose of sedation can improve patient tolerance and hence safety without additional side effects. Similar findings have reported in gastroenterology and surgery units, where moderate sedation with analgesia not only improved the patient comfort and procedural cooperation but also reduced the peri-procedural anxiety, better patient satisfaction and decreased risk of procedure interruption.

Ketorolac tromethamine (Toradol) is a highly effective nonsteroidal anti-inflammatory drug (NSAID) with potent analgesic action without inducing respiratory depression. When administered intravenously prior to bronchoscopy, ketorolac may reduce pain, improve comfort, and maintain cardiovascular stability. It has a rapid onset and is generally safe to combine with sedatives such as midazolam. To ensure patient safety, individuals with known contraindications to NSAIDs, including bronchial asthma, are excluded from the present study.

This study therefore aims to compare the effects of midazolam alone versus midazolam combined with ketorolac on patient comfort, sedation quality, and safety during flexible bronchoscopy. The results may assist in designing a more effective and patient-friendly sedation strategy for bronchoscopy in Pakistan.

DETAILED DESCRIPTION:
Flexible bronchoscopy has emerged as a cornerstone in the evaluation and management of respiratory diseases, providing clinicians with the ability to directly visualize the tracheobronchial tree and perform a wide array of diagnostic and therapeutic procedures. Its applications include bronchoalveolar lavage for cytological and microbiological analysis, endobronchial tissue biopsy for histopathological assessment, and removal of foreign bodies or secretions obstructing the airway. Despite its widespread use and clinical importance, flexible bronchoscopy remains a procedure that can cause significant discomfort and anxiety for patients. The manipulation of the airway often triggers coughing, dyspnea, hypoxia, and pain, which may lead to excessive movement, impaired cooperation, and in some cases, premature termination of the procedure. These challenges can compromise both patient safety and the accuracy of diagnostic outcomes.

To mitigate these issues, sedation and analgesia are routinely employed to improve procedural tolerance. Effective sedation reduces anxiety, suppresses involuntary airway reflexes, and shortens procedure duration, all while maintaining patient safety. The ideal sedative agent for bronchoscopy should achieve a balance between adequate sedation and rapid recovery, allowing for procedural efficiency, patient comfort, and optimal diagnostic yield. However, the use of sedative agents is not without risk. Dose-dependent complications, such as bradycardia, hypotension, respiratory depression, and hypoxia, may occur and can necessitate interruption or termination of the procedure. Furthermore, the use of topical anesthetics like lignocaine at higher doses carries the potential for serious adverse effects including seizures and cardiac arrhythmias.

Research in both pulmonary medicine and other procedural disciplines, such as gastroenterology and surgery, has demonstrated that combining analgesics with sedative agents can enhance patient comfort and procedural cooperation while minimizing complications. Moderate sedation combined with analgesia has been associated with reduced peri-procedural anxiety, improved patient satisfaction, decreased risk of procedural interruption, and overall better procedural outcomes. This approach leverages the synergistic effects of sedatives and analgesics to provide a safer and more tolerable procedural experience.

Ketorolac tromethamine (Toradol) is a potent nonsteroidal anti-inflammatory drug with strong analgesic properties that does not induce respiratory depression, making it an attractive option for procedural analgesia. Intravenous administration of ketorolac prior to bronchoscopy has been shown to improve patient comfort, reduce pain, and maintain cardiovascular stability. Its rapid onset and favorable safety profile allow for safe co-administration with sedative agents such as midazolam. To ensure patient safety, individuals with contraindications to NSAIDs, including those with bronchial asthma, are excluded from this study.

The primary objective of this study is to evaluate and compare the effects of midazolam alone versus midazolam combined with ketorolac on patient comfort, sedation quality, and safety during flexible bronchoscopy. Secondary objectives include assessing procedural tolerance, incidence of adverse events, hemodynamic stability, and overall patient satisfaction. By systematically investigating the benefits of combining analgesia with sedation, this study aims to inform the development of evidence-based sedation protocols that optimize patient comfort, safety, and procedural efficiency.

The findings from this research have the potential to impact clinical practice significantly, particularly in resource-limited settings like Pakistan, where optimizing procedural sedation strategies can enhance patient experience, improve diagnostic accuracy, and minimize procedural complications. This study addresses a critical gap in the literature regarding the synergistic use of sedatives and analgesics during bronchoscopy and may provide guidance for safe and effective sedation practices that can be widely adopted in clinical respiratory medicine.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-75 years. Patients undergoing flexible bronchoscopy. ASA physical status I-III. Patients able to provide informed written consent.

-

Exclusion Criteria:

* History of bronchial asthma or NSAID-exacerbated respiratory disease (NERD). Known hypersensitivity or contraindication to midazolam or NSAIDs (e.g., ketorolac).

Coagulopathy or platelet count < 70,000/µL. Active peptic ulcer disease or diagnosed bleeding disorder. Severe renal impairment CKD grade 3 or 4 with eGFR <50ml/min or hepatic failure.

Chronic opioid use or benzodiazepine dependency. Unstable cardiorespiratory status (e.g., respiratory failure or requiring high-flow oxygen).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of sedation-related adverse events. | During the procedure and within 30 mints after bronchoscopy.
  Sedation-related adverse events including hypoxia, hypotension, bradycardia, need for airway intervention, or premature termination of procedure will be recorded and compared between groups.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang CP, Cherng CH, Wong CS, Ho ST. Effects of intravenous ketorolac and fentanyl combined with midazolam on analgesia and side effects during extracorporeal shock wave lithotripsy. Acta Anaesthesiol Sin. 2002 Mar;40(1):9-12. PMID 11989050

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT07352059/Prot_SAP_000.pdf